CLINICAL TRIAL: NCT00131963
Title: A Pharmacogenomics Study for Breast Cancer Patients Undergoing Adjuvant Chemotherapy With Doxorubicin (A)/Cyclophosphamide ©) and/or Weekly Paclitaxel
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00014267; DUMC-4522-04-1-R1 (Other: Duke IRB); CDR0000438673 (Other: National Cancer Institute)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: stage One A (IA) breast cancer; stage Two (II) breast cancer; stage Three A (IIIA) breast cancer; stage Three B(IIIB) breast cancer; stage Three C(IIIC) breast cancer; stage One B (IB) breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from blood samples taken at the first cycle of Doxorubicin and/or Paclitaxel to analyze certain genes that may predict the severity of side-effects that may be experienced with chemotherapy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regimen 1: Patients receive doxorubicin IV over 10 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin
- Regimen 2: Patients receive doxorubicin and cyclophosphamide as in regimen 1. Patients then receive paclitaxel IV over 1 hour once weekly for 12 weeks.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin; Drug: paclitaxel

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan
Drug: doxorubicin — Given IV
  Other Names: adriamycin
Drug: paclitaxel — Given IV
  Other Names: taxol
  Groups: Regimen 2

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well doxorubicin, cyclophosphamide, and/or paclitaxel work in treating women with nonmetastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pharmacogenomics of adjuvant chemotherapy comprising doxorubicin and cyclophosphamide and/or paclitaxel in women with nonmetastatic invasive breast cancer.
* Determine treatment-induced myelosuppression (e.g., neutropenia) in patients treated with adjuvant doxorubicin and cyclophosphamide who have polymorphisms in drug activation and metabolism genes.
* Correlate the incidence of peripheral neuropathy with pharmacogenomic analysis in patients treated with paclitaxel.

Secondary

* Determine response (i.e., relapse in the adjuvant setting) during a 10-year follow-up period in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients receive treatment on The Cancer and Leukemia Group B study(CALGB) CALGB-40101 OR are assigned to receive 1 of 2 treatment regimens on this study.

* Regimen 1: Patients receive doxorubicin IV over 10 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.
* Regimen 2: Patients receive doxorubicin and cyclophosphamide as in regimen 1. Patients then receive paclitaxel IV over 1 hour once weekly for 12 weeks.

After completion of study treatment, patients are followed at 3, 6, and 12 months and then annually for up to 10 years.

PROJECTED ACCRUAL: A total of 500 patients (300 treated with doxorubicin and cyclophosphamide and 200 treated with paclitaxel) will be accrued for this study within 3-4 years.

ELIGIBILITY:
Eligibility Criteria

* Histologically confirmed invasive breast cancer
* node negative stage > T1c or T1b with poor prognostic features (high grade, Her2/neu FISH positive, ER negative) or stage 2 (T2, N0) or
* enrolled on CALGB 40101, CALGB 49909, or the National Cancer Institute of Canada study MA-21 or
* any node positive patient or locally advanced undergoing neoadjuvant chemotherapy with either AC or paclitaxel
* Age greater than or equal to 18 years.
* >/=2 weeks from major surgery (wide excision / lumpectomy / mastectomy)
* No evidence of systemic metastasis
* Undergoing adjuvant treatment with standard dose AC or AC followed by weekly Paclitaxel at 80mg/m2
* Adequate bone marrow, hepatic and renal functions (absolute neutrophil count >1,500/ μl, platelet count > 100,000/ μl, serum creatinine <2.0 mg/dl, total Bilirubin <2.0 x the upper limit of normal (ULN)
* Ability to answer and understand study surveillance questionnaires
* No concurrent drug therapy (within 2 weeks) with agents that are known inducers or inhibitors of Cytochrome P450 (CYP450).

Exclusion Criteria

* Other anticancer cytotoxic or endocrine therapy, immunotherapy, or biologic response modifiers,Study Drugs or other concomitant medications known to cause myelosuppression especially neutropenia and neuropathy
* Eastern Cooperative Oncology Group Performance Status(ECOG) functional status > 2.
* Serious co-morbidities including poorly controlled diabetes mellitus, ischaemic heart disease,uncontrolled hypertension or active infection.
* Pregnancy
* Use of growth factor during cycle 1 of chemotherapy (AC) under pharmacokinetic evaluation
* Grade >/=2 peripheral neuropathy symptoms based on National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE) Scale. Exception: a chronic neurologic disorder will be reviewed on a case by case basis by the study PI.
* Prior treatment with weekly paclitaxelDISEASE CHARACTERISTICS:

  * Histologically confirmed invasive breast cancer, meeting 1 of the following criteria:

    * Node negative disease AND meets 1 of the following stage criteria:

      * Primary tumor > T1c
      * Primary tumor > T1b AND poor prognostic features, defined as the following:

        * High-grade disease
        * Human Epidermal Growth Factor Receptor 2 (HER2)/neu-positive disease by fluorescence in situ hybridization
        * Estrogen receptor-negative disease
      * Stage II disease (T2, N0)
    * Node positive nonmetastatic disease
    * Locally advanced disease AND receiving neoadjuvant chemotherapy comprising doxorubicin and cyclophosphamide OR paclitaxel
    * Enrolled in clinical trial CALGB-40101
  * No evidence of systemic metastasis
  * Hormone receptor status:

    * Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the breast cancer oncology clinics.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2003-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Treatment-induced myelosuppression (e.g., neutropenia) | 12 months
Incidence of peripheral neuropathy | 12 month

SECONDARY OUTCOMES:
Response (relapse in adjuvant setting) for 10 years after completion of study treatment | Ten years

CONTACTS AND LOCATIONS:
Overall Officials: Paul K. Marcom, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States